CLINICAL TRIAL: NCT00708214
Title: A Phase II Study of BIBW 2992 Administration in Patients With Hormone Refractory Metastatic Breast Cancer
Brief Title: BIBW 2992 and Letrozole in Hormonoresistant Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 1200.5; 2006-002814-37 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-06-30; First posted 2008-07-02 (Estimated); Results first posted 2013-11-19 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-10

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Afatinib; Letrozole

ARMS (2):
- BIBW 2992 (Experimental): To study BIBW 2992 in association with letrozole in hormonoresistant metastatic breast cancer
  Interventions: Drug: BIBW 2992; Drug: Letrozole
- Letrozole (Other): Hormonotherapy for metastatic breast cancer
  Interventions: Drug: BIBW 2992; Drug: Letrozole

INTERVENTIONS:
Drug: BIBW 2992 — BIBW 2992 at high and medium dosages
  Arms: BIBW 2992
Drug: BIBW 2992 — BIBW 2992 at high and medium dosages
  Arms: Letrozole
Drug: Letrozole — Letrozole at standard dosage
  Arms: BIBW 2992
Drug: Letrozole — Letrozole at standard dosage
  Arms: Letrozole

SUMMARY:
Progression-free rate after 16 weeks of BIBW 2992 administration in association with letrozole

ELIGIBILITY:
Inclusion criteria:

* Female patients with histologically proven breast adenocarcinoma
* Presence of metastatic disease No more than 2 prior chemotherapy regimens for metastatic disease, which could include trastuzumab Patients must currently be on letrozole and developed acquired resistance as defined by disease progression on letrozole following previous response (partial response or better, stable disease superior or equal to 24 weeks)

Diagnosis of disease progression inferior or equal to 6 weeks prior to trial entrydefined as:

1. Increase in the number of bone lesions on bone scan or on MRI AND/OR
2. Increased pain in an area of known bony metastasis AND superior or equal to 2 serial elevations in CA 15.3 AND/OR
3. Progression according to RECIST criteria on CT scan, MRI, or x-ray Patients must have documented menopause confirmed by estradiol level inferior to 11 pg/ml

Exclusion criteria:

* Premenopausal patients
* Rapidly progressive disease in major organs (i.e. lymphangitic spread in the lung and/or bulky liver metastasis) Patient with brain metastasis Significant cardiovascular diseases Previous treatment with an EGFR and/or HER-2 inhibiting drug(patients who received trastuzumab with chemotherapy but not with letrozole can be enrolled)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-01; Primary Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (5):
- France (5):
  - 1200.5.3306A Boehringer Ingelheim Investigational Site, Caen
  - 1200.5.3304A Boehringer Ingelheim Investigational Site, Nice
  - 1200.5.3301A Boehringer Ingelheim Investigational Site, Paris
  - 1200.5.3305A Boehringer Ingelheim Investigational Site, Paris
  - 1200.5.3302A Boehringer Ingelheim Investigational Site, Saint-Cloud

REFERENCES:
- [Derived] Gunzer K, Joly F, Ferrero JM, Gligorov J, de Mont-Serrat H, Uttenreuther-Fischer M, Pelling K, Wind S, Bousquet G, Misset JL. A phase II study of afatinib, an irreversible ErbB family blocker, added to letrozole in patients with estrogen receptor-positive hormone-refractory metastatic breast cancer progressing on letrozole. Springerplus. 2016 Jan 19;5:45. doi: 10.1186/s40064-015-1601-7. eCollection 2016. PMID 26835225

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: According to the protocol the starting dose of Afatinib was 50mg/day. This dose was reduced according to the protocol to first 40mg/day and then to 30mg/day due to skin toxicity.
Groups:
- Afatinib 50 mg With Letrozole: Patients received continuous daily dosing with Afatinib 50 mg therapy with letrozole 2.5 mg over 28-day treatment cycles until further disease progression.
- Afatinib 40 mg With Letrozole: Patients received continuous daily dosing with Afatinib 40 mg therapy with letrozole 2.5 mg over 28-day treatment cycles until further disease progression.
- Afatinib 30 mg With Letrozole: Patients received continuous daily dosing with Afatinib 30 mg therapy with letrozole 2.5 mg over 28-day treatment cycles until further disease progression.
Period: Overall Study
Arm/Group | Afatinib 50 mg With Letrozole | Afatinib 40 mg With Letrozole | Afatinib 30 mg With Letrozole
Started | 7 | 13 | 8
Completed | 0 (On treatment at analysis cut-off date (04 Jan 2010)) | 0 (On treatment at analysis cut-off date (04 Jan 2010)) | 0 (On treatment at analysis cut-off date (04 Jan 2010))
Not Completed | 7 | 13 | 8
Not completed — Other Adverse Event | 3 | 6 | 2
Not completed — Other | 0 | 1 | 1
Not completed — Progressive Disease | 4 | 6 | 5

BASELINE CHARACTERISTICS:
Population: Treated set (TS). TS consisted of all patients who were dispensed study medication and have taken at least 1 dose of Afatinib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Afatinib 50 mg With Letrozole | Afatinib 40 mg With Letrozole | Afatinib 30 mg With Letrozole | Total
Number analyzed (Participants) | 7 | 13 | 8 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (14.7) | 64.8 (7.2) | 58.5 (9.0) | 62.5 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 8 | 28
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Progression Free Participants After 16 Weeks of Treatment
Description: Progression was defined according to 1 of the following criteria: New bone lesion(s) on bone scan or on magnetic resonance imaging; Progression or occurrence of new lesion(s) according to the Response Evaluation Criteria In Solid Tumours version 1.0 (RECIST); an increase in tumour marker CA 15.3 of more than 20 percent,compared with baseline, at 2 consecutive examinations; occurrence of disease-related skeletal events. If a patient did not fulfil any criteria and was withdrawn because of clinical deterioration amounting to PD according to the Investigator, they were considered as having PD.
Time Frame: 16 weeks
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Afatinib 50 mg With Letrozole | Afatinib 40 mg With Letrozole | Afatinib 30 mg With Letrozole
Number analyzed (Participants) | 7 | 13 | 8
Percentage of participants | 28.57 [3.67 to 70.96] | 0.00 [0.00 to 24.71] | 25.00 [3.19 to 65.09]

2. Secondary Outcome: Number of Participants With Confirmed Objective Response (OR)
Description: OR was defined as complete response (CR) or partial response (PR) and was assessed according to RECIST criteria regardless of treatment status.
Time Frame: Baseline till progression
Population: TS
Measure: Number; unit: Participants
Arm/Group | Afatinib 50 mg With Letrozole | Afatinib 40 mg With Letrozole | Afatinib 30 mg With Letrozole
Number analyzed (Participants) | 7 | 13 | 8
Participants | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Clinical Benefit (CB)
Description: CB was defined as CR, PR or stable disease (SD) and was assessed according to RECIST criteria regardless of treatment status.
Time Frame: 16 weeks and 24 weeks
Population: TS
Measure: Number; unit: Participants
Arm/Group | Afatinib 50 mg With Letrozole | Afatinib 40 mg With Letrozole | Afatinib 30 mg With Letrozole
Number analyzed (Participants) | 7 | 13 | 8
Participants
  Participants with CB at 16 weeks | 2 | 2 | 2
  Participants with CB at 24 weeks | 2 | 0 | 2

4. Secondary Outcome: Time to RECIST Tumour Reponse
Description: The time to OR was the duration from the first treatment to the time when the measurement criteria for CR and/or PR were met according to RECIST criteria.
Time Frame: Baseline till progression
Population: TS. Median time to RECIST tumour response was not calculable as there was no OR observed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Afatinib 50 mg With Letrozole | Afatinib 40 mg With Letrozole | Afatinib 30 mg With Letrozole
Number analyzed (Participants) | 7 | 13 | 8
days | NA [NA to NA] — Median time to RECIST tumour response was not calculable as there was no OR observed. | NA [NA to NA] — Median time to RECIST tumour response was not calculable as there was no OR observed. | NA [NA to NA] — Median time to RECIST tumour response was not calculable as there was no OR observed.

5. Secondary Outcome: Duration of Confirmed OR
Description: Duration of confirmed OR is measured from the time of first OR to the time of progression or death (or date of censoring for progression free survival).
Time Frame: First occurence or OR till progression or death
Population: TS. Median duration of RECIST tumour response was not calculable as there was no OR observed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Afatinib 50 mg With Letrozole | Afatinib 40 mg With Letrozole | Afatinib 30 mg With Letrozole
Number analyzed (Participants) | 7 | 13 | 8
days | NA [NA to NA] — Median duration of RECIST tumour response was not calculable as there was no OR observed. | NA [NA to NA] — Median duration of RECIST tumour response was not calculable as there was no OR observed. | NA [NA to NA] — Median duration of RECIST tumour response was not calculable as there was no OR observed.

6. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the first treatment to the occurrence of tumour progression or death, whichever came first. Progression was assessed according to RECIST criteria.
Time Frame: Baseline till progression, death or data cut-off (04 Jan 2010)
Population: TS
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Afatinib 50 mg With Letrozole | Afatinib 40 mg With Letrozole | Afatinib 30 mg With Letrozole
Number analyzed (Participants) | 7 | 13 | 8
days | 60.0 [51.0 to 443.0] | 107.0 [44.0 to 163.0] | 79.0 [21.0 to 230.0]

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first treatment to death.
Time Frame: Baseline till progression, death or data cut-off
Population: TS. Estimation of median time to death was not feasible, due to the small number of patients who died during the trial.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Afatinib 50 mg With Letrozole | Afatinib 40 mg With Letrozole | Afatinib 30 mg With Letrozole
Number analyzed (Participants) | 7 | 13 | 8
days | NA [208.0 to NA] — Estimation of median time to death was not feasible, due to the small number of patients who died during the trial. | NA [288.0 to NA] — Estimation of median time to death was not feasible, due to the small number of patients who died during the trial. | NA [137.0 to NA] — Estimation of median time to death was not feasible, due to the small number of patients who died during the trial.

8. Secondary Outcome: Area Under Curve of Afatinib Over a Uniform Dosing Interval Tau at Steady State (AUCtau,ss)
Description: AUCtau,ss represents the area under the concentration curve of afatinib in plasma over a uniform dosing interval tau at steady state.
Time Frame: 0.05 hours (h) before dosing and 2h, 4h, 6h, 8h and 24h after dosing
Population: Data were particularly sparse for the 50 mg starting dose group and were not summarised.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Afatinib 40 mg: Patients received continuous daily dosing with Afatinib 40 mg therapy with letrozole 2.5 mg over 28-day treatment cycles until further disease progression.
- Afatinib 30 mg: Patients received continuous daily dosing with Afatinib 30 mg therapy with letrozole 2.5 mg over 28-day treatment cycles until further disease progression.
Arm/Group | Afatinib 40 mg | Afatinib 30 mg
Number analyzed (Participants) | 4 | 5
ng*h/mL | 660 (41.3) | 579 (62.8)

9. Secondary Outcome: Maximum Concentration of Afatinib in Plasma at Steady State (Cmax,ss)
Description: Cmax,ss represents the maximum measured concentration of afatinib in plasma at steady state.
Time Frame: 0.05 hours (h) before dosing and 2h, 4h, 6h, 8h and 24h after dosing
Population: Data were particularly sparse for the 50 mg starting dose group and were not summarised.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Afatinib 40 mg | Afatinib 30 mg
Number analyzed (Participants) | 4 | 5
ng/mL | 43.8 (42.0) | 33.9 (79.4)

10. Secondary Outcome: Pre-dose Concentration of Afatinib in Plasma at Steady State on Day 57 (Cpre,ss,57)
Description: Cpre,ss,57 represents the pre-dose concentration of afatinib in plasma at steady state on day 57.
Time Frame: Day 57
Population: Data were particularly sparse for the 50 mg starting dose group and were not summarised.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Afatinib 40 mg | Afatinib 30 mg
Number analyzed (Participants) | 5 | 8
ng/mL | 21.4 (42.3) | 15.8 (42.1)

11. Secondary Outcome: Pre-dose Concentration of Afatinib in Plasma at Steady Stateon Day 85 (Cpre,ss,85)
Description: Cpre,ss,85 represents the pre-dose concentration of afatinib in plasma at steady state on day 85.
Time Frame: Day 85
Population: Data were particularly sparse for the 50 mg starting dose group and were not summarised.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Afatinib 40 mg | Afatinib 30 mg
Number analyzed (Participants) | 4 | 5
ng/mL | 16.9 (55.7) | 17.3 (46.5)

12. Secondary Outcome: Time From Dosing to the Maximum Concentration of Afatinib in Plasma at Steady State (Tmax,ss)
Description: tmax,ss represents the time from dosing to the maximum concentration of afatinib in plasma at steady state
Time Frame: 0.05 hours (h) before dosing and 2h, 4h, 6h, 8h and 24h after dosing
Population: Data were particularly sparse for the 50 mg starting dose group and were not summarised.
Measure: Median (Full Range); unit: hours
Arm/Group | Afatinib 40 mg | Afatinib 30 mg
Number analyzed (Participants) | 4 | 5
hours | 2.00 (2.00-4.00) [2.00 to 4.00] | 4.00 (0.917-7.67) [0.917 to 7.67]

13. Secondary Outcome: Area Under Curve of Letrozole Over a Uniform Dosing Interval Tau at Steady State (AUCtau,ss)
Description: AUC0-tau,ss represents the area under the concentration curve of letrozole in plasma over a uniform dosing interval tau at steady state.
Time Frame: 0.05 hours (h) before dosing and 2h, 4h, 6h, 8h and 24h after dosing
Population: Analysis of all treatment arms combined, as Letrozole dose was the same in all arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Afatinib Overall, With Letrozole 2.5 mg: Patients received continuous daily dosing with Afatinib 30, 40 or 50 mg therapy with letrozole 2.5 mg over 28-day treatment cycles until further disease progression.
Arm/Group | Afatinib Overall, With Letrozole 2.5 mg
Number analyzed (Participants) | 10
ng*h/mL | 2420 (76.2)

14. Secondary Outcome: Maximum Concentration of Letrozole in Plasma at Steady State (Cmax,ss)
Description: Cmax,ss represents the maximum measured concentration of letrozole in plasma at steady state.
Time Frame: 0.05 hours (h) before dosing and 2h, 4h, 6h, 8h and 24h after dosing
Population: Analysis of all treatment arms combined, as Letrozole dose was the same in all arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Afatinib Overall, With Letrozole 2.5mg: Patients received continuous daily dosing with Afatinib 30, 40 or 50 mg therapy with letrozole 2.5 mg over 28-day treatment cycles until further disease progression.
Arm/Group | Afatinib Overall, With Letrozole 2.5mg
Number analyzed (Participants) | 10
ng/mL | 135 (70.0)

15. Secondary Outcome: Time From Dosing to the Maximum Concentration of Letrozole in Plasma at Steady State (Tmax,ss)
Description: tmax,ss represents the time from dosing to the maximum concentration of letrozole in plasma at steady state.
Time Frame: 0.05 hours (h) before dosing and 2h, 4h, 6h, 8h and 24h after dosing
Population: Analysis of all treatment arms combined, as Letrozole dose was the same in all arms.
Measure: Median (Full Range); unit: hours
Arm/Group | Afatinib Overall, With Letrozole 2.5mg
Number analyzed (Participants) | 10
hours | 1.00 [0.917 to 23.8]

16. Secondary Outcome: Change From Baseline in Ca15.3
Description: Change from baseline in Ca15.3 tumor marker levels
Time Frame: baseline and day 29
Population: Analysis of all treatment arms combined for tumor marker analysis.
Measure: Median (Full Range); unit: percentage of baseline level
Groups:
- Afatinib Overall: Patients received continuous daily dosing with Afatinib 30, 40 or 50 mg therapy with letrozole 2.5 mg over 28-day treatment cycles until further disease progression.
Arm/Group | Afatinib Overall
Number analyzed (Participants) | 21
percentage of baseline level | -4.35 [-28.4 to 41.8]

17. Secondary Outcome: Best Change From Baseline in ECOG Performance Status
Description: Best change from baseline in ECOG (Eastern Cooperative Oncology Group) performance status. ECOG is measured as score between 0 (fully active) and 5 (dead). Improvement is a decrease in ECOG score from baseline of at least 1. Deterioration is an increase in ECOG score from baseline of at least 1
Time Frame: baseline till end of treatment
Measure: Number; unit: participants
Arm/Group | Afatinib Overall
Number analyzed (Participants) | 28
participants
  Improved | 4
  Deteriorated | 6
  Unchanged | 16
  Not done | 2

ADVERSE EVENTS:
Time Frame: First administration of trial medication until 28 days after last administration of trial medication
Arm/Group | Afatinib 50 mg With Letrozole | Afatinib 40 mg With Letrozole | Afatinib 30 mg With Letrozole
Serious Adverse Events (participants affected / at risk) | 1/7 | 3/13 | 5/8
Other Adverse Events (participants affected / at risk) | 7/7 | 13/13 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 50 mg With Letrozole (N=7) | Afatinib 40 mg With Letrozole (N=13) | Afatinib 30 mg With Letrozole (N=8)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1 | 0
Obstruction (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 1 | 0
Post precedural sepsis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 50 mg With Letrozole (N=7) | Afatinib 40 mg With Letrozole (N=13) | Afatinib 30 mg With Letrozole (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 2 | 2 | 2
Dry eye (Eye disorders) | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 1
Eyelid disorder (Eye disorders) | 1 | 0 | 0
Eyelid irritation (Eye disorders) | 1 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 1
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 1 | 2
Cheilitis (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 12 | 7
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 4 | 3
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 3 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0
Asthenia (General disorders) | 4 | 8 | 4
Catheter site inflammation (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Cyst (General disorders) | 0 | 0 | 1
Facial pain (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Hypothermia (General disorders) | 1 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 1
Mucosal inflammation (General disorders) | 5 | 3 | 2
Oedema (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Pain (General disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 0
Food allergy (Immune system disorders) | 1 | 0 | 0
Cystitis (Infections and infestations) | 2 | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 2
Hordeolum (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0
Paronychia (Infections and infestations) | 1 | 1 | 2
Rhinitis (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 4 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Muscle spasm (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 4 | 2
Epiduritis (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 4 | 0 | 2
Neuralgia (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 3 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0
Genital burning sensation (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 1 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 5 | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 5 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 4 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 5 | 6
Skin fissures (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.